CLINICAL TRIAL: NCT05762419
Title: A Feasibility Study Examining the Use of Non-Invasive Focused Ultrasound (FUS) With Oral Etoposide Administration in Children With Progressive Diffuse Midline Glioma (DMG)
Brief Title: FUS Etoposide for DMG
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Focused Ultrasound Foundation (Other)
Responsible Party: Principal Investigator, Stergios Zacharoulis, Herbert and Florence Irving Associate Professor of Pediatric Neuro-Oncology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAU1228
Record Dates: First submitted 2023-02-06; First posted 2023-03-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Diffuse Midline Glioma, H3 K27M-Mutant
Keywords: bood brain barrier; diffuse midline glioma; focused ultrasound; pontine glioma; thalamic glioma; DIPG; DMG; Glioma; Brain Diseases; Nervous System Neoplasms; Central Nervous System Neoplasm; Etoposide; Diffuse Intrinsic Pontine Glioma; Brain Neoplasms
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Glioma; Brain Diseases; Nervous System Neoplasms; Central Nervous System Neoplasms; Brain Neoplasms | interventions — Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Focused ultrasound using oral etoposide (Experimental): All patients enrolled in the study will be treated with oral etoposide after receiving focused ultrasound (FUS) treatment with microbubbles and neuro-navigator-controlled sonication.
  Interventions: Drug: Etoposide; Oral, 50 Mg; Device: Focused ultrasound with neuro-navigator-controlled sonication

INTERVENTIONS:
Drug: Etoposide; Oral, 50 Mg — Subjects will receive focused ultrasound sonication followed by once daily oral etoposide (50mg/m^2/dose). Oral etoposide will be taken every day for 21 days, followed by one week of rest. For the first cycle, etoposide will be administered immediately following confirming of the blood brain barrier opening through contrast magnetic resonance imaging (MRI) which will occur within 4 hours of the focused ultrasound procedure. For subsequent cycles, etoposide will be administered immediately following the focused ultrasound procedure. Subjects may continue for a maximum of 4 cycles.
  Other Names: Etoposide phosphate
Device: Focused ultrasound with neuro-navigator-controlled sonication — Focused ultrasound sonication will be performed a maximum of three times a week for two weeks with two weeks of rest.

SUMMARY:
The blood brain barrier (BBB) prevents some drugs from successfully reaching the target tumor. Focused Ultrasound (FUS) using microbubbles and neuro-navigator controlled sonication is a non-invasive method of temporarily opening up the blood brain barrier to allow a greater concentration of the drug to reach into the brain tumor. This may improve response and may also reduce system side effects in the patient.

The primary purpose of this study is to evaluate the feasibility of safely opening the blood brain barrier in children with progressive diffuse midline gliomas (DMG) treated with oral etoposide using focused ultrasound with microbubbles and neuro-navigator-controlled sonication.

For the purpose of the study, the investigators will be opening up the blood brain barrier temporarily in one or two locations around the tumor using the non-invasive focused ultrasound technology, and administrating oral etoposide in children with progressive diffuse midline glioma.

DETAILED DESCRIPTION:
Diffuse midline gliomas constitute 10% of all pediatric central nervous system (CNS) tumors. Subjects with Diffuse Intrinsic Pontine Gliomas (DIPG) have a poor prognosis with a median survival that is usually reported to be 9 months, and nearly 90% of children die within 18 months from diagnosis. The mainstay of treatment is radiation to the primary tumor site. Surgical resection does not influence the outcome and is often not feasible in this part of the central nervous system.

Many promising drugs for central nervous system disorders have failed to attain clinical success due to an intact blood brain barrier, limiting their access from the systemic circulation into the brain. Systemic administration of high doses may increase delivery to the brain, but this approach risks significant side effects and systemic toxicities. Direct delivery of the drugs to the brain by injection into the parenchyma bypasses the blood brain barrier; however, drug distribution from the site of injection tends to be limited.

The technique of using focused ultrasound with microbubbles and neuro-navigator-controlled sonication can temporarily open up the blood brain barrier and allow for a greater concentration of drug to reach the tumor, thus potentially improving response in patients.

With the current study, the investigators are planning to evaluate the safety and feasibility of using focused ultrasound and open-space neuronavigator-controlled sonication to open one to two tumor sites. For the purpose of the study, investigators will be administrating oral etoposide in children with progressive diffuse midline glioma. This drug has a known toxicity profile, dose, and well-documented efficacy against many metastatic cancers. Successful opening and closing of the blood brain barrier will be confirmed with periodic magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Ages 4 - 21 years
* Radiological diagnosis of Diffuse Midline Glioma with tumor involving the pons (intrinsic, pontine based infiltrative lesion; hypointense on T1 weighted images (T1WIs) and hyperintense in T2 sequences, with mass effect on the adjacent structures and occupying at least 50% of the pons), thalami, and/or histological confirmation of H3K27M mutation of pontine or thalamic glioma. Subjects must have evidence of clinical and/or radiographic progression of disease.
* Lansky performance status score of at least 60 for subjects 16 years of age or younger.
* Karnofsky performance status of at least 60 for subjects greater than 16 years of age
* Organ Function:

  * Adequate hematologic function defined as:

    * Peripheral absolute neutrophil count ≥ 1,500/µL
    * Platelet count ≥ 100,000/µL
    * Partial thromboplastin time (PTT) and activated partial thromboplastin time (APTT): within normal institutional limits
  * Adequate renal function defined as:

    * Potassium and magnesium levels within institutional limits
    * Serum creatinine below the institutional upper limit of normal (ULN) for age and gender, or creatinine clearance: ≥ 60 mL/min/1.73m2
  * Adequate hepatic function defined as:

    * Total bilirubin below the institutional ULN for age
    * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 × institutional ULN
* Prior Therapy:

  * Subjects must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment.
  * Cytotoxic chemotherapy or anti-cancer agents known to be myelosuppressive: at least 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy.
  * Anti-cancer agents not known to be myelosuppressive: at least 7 days must have elapsed from last dose of agent.
  * Antibodies: at least 21 days must have elapsed from infusion of last dose of antibody.
  * Interleukins, interferons, and cytokines: at least 21 days must have elapsed since the completion of interleukins, interferon, or cytokines.
  * Stem cell infusions: at least 42 days must have elapsed after completion of an autologous stem cell infusion, and at least 84 days must have elapsed after completion of an allogeneic stem cell infusion.
  * Cellular therapy: at least 42 days must have elapsed since the completion of any type of cellular therapy
  * Radiotherapy (XRT): at least 1 month must have elapsed after local XRT.
  * Subjects must be on a stable or decreasing dose of steroids, as well as stable dose of anti-seizure medication for at least 1 week.
* Subject able to give consent

Exclusion Criteria:

* Subjects that have previously received etoposide therapy
* Subjects unable to tolerate study procedures and/or anesthesia based on the opinion of the principal investigator
* Uncontrolled seizure disorder
* Pregnancy or Breast-Feeding: pregnant or breast-feeding women will not be entered on this study, since there is yet no available information regarding human fetal or teratogenic toxicities; a pregnancy test must be obtained in girls who are post-menarchal. Males with female partners of reproductive potential or females of reproductive potential may not participate unless they have agreed to use two effective methods of birth control- including a medically accepted barrier method of contraception (e.g., a male or female condom) for the entire period in which they are receiving protocol therapy and for at least 1 month following their last study treatment requirement. Abstinence is an acceptable method of birth control. Women of childbearing potential will be provided a routine quantitative beta-human chorionic gonadotropin (B-hCG) test during the pre-study phase, prior to enrollment and each cycle.
* Concomitant medications: subjects who are currently receiving another investigational drug or other anti-cancer agents are not eligible.
* Screening EKG with a QTc > 450 msec.
* Subjects with evidence of active systemic infection
* Subjects with a documented allergy to compounds of similar chemical or biologic composition to etoposide or gadolinium compounds
* Subjects with implanted metallic or electrical devices
* Subjects with uncontrollable hypertension
* Subjects with a documented bleeding disorder
* Subjects with history of structural cardiac anomalies or arrhythmias
* Subjects with history of unprovoked stroke or signs of stroke in the area of FUS target
* Subjects with SARS-CoV-2 infection requiring hospitalization in the past month and requires anticoagulation as per the Columbia University Irving Medical Center (CUIMC) institutional "Anticoagulation for COVID-19 Positive Pediatric Inpatients" guidelines (See Appendix B)
* Subjects with coagulopathy or under anticoagulant therapy.
* Subjects with signs of impending herniation or an acute or previous intratumoral hemorrhage
* Subjects with spinal cord diffuse midline glioma
* Subjects receiving a drug where CNS toxicity is reasonably suspected

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of total adverse events | Up to 90 days after the end of the last focused ultrasound treatment
  This is to evaluate the safety of using focused ultrasound to open the blood brain barrier at one or two sites for administration of etoposide in children with progressive diffuse midline glioma. Safety will be assessed by adverse events as per the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (including abnormalities from physical and neurologic examinations, laboratory values, and radiographic results).
Number of patients with successful opening of the blood brain barrier | Treatment will consist of up to 4 cycles, each lasting 28 days. During the first 2 weeks of each cycle, subjects will receive FUS therapy for a maximum of 3 times per week, concurrent with etoposide.
  This is to evaluate the feasibility of using FUS to open the blood brain barrier at one or two sites for administration of etoposide in children with progressive diffuse midline glioma. The study defines feasibility as successful opening of the blood brain barrier.

SECONDARY OUTCOMES:
3-month Progression Free Survival (PFS3) | Up to 3 months after last focused ultrasound treatment
  Progression Free Survival is defined as the duration of the time from the start of focused ultrasound treatment to time of progression or death from any cause, whichever occurs first. Patient's vitality status will be monitored with a monthly follow-up phone call for 3 months post-treatment.
3-month Overall Survival (OS3) | Up to 3 months after last focused ultrasound treatment
  Overall survival is defined as the duration of time from the start of focused ultrasound treatment to death from any cause. Overall survival will be measured by follow-up with a study participant every 3-6 months until death for any reason. Patient's vitality status will be monitored with a monthly follow-up phone call for 3 months post-treatment.
Blood brain barrier/Tumor imaging changes | Up to 90 days after the end of the last focused ultrasound treatment
  MRI and other radiological evidence to show successful BBB opening and closing
Number of severe or serious adverse events | Up to 90 days after the last focused ultrasound treatment
  All severe adverse events (SAEs), and adverse events (AEs), grade 3 and higher (except for thrombocytopenia which will include grade 2) will be collected and reported on each patient over the course of their treatment, according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. All SAEs and any AEs grade 3 and higher (except for thrombocytopenia which will include grade 2) will be tallied.

CONTACTS AND LOCATIONS:
Overall Officials: Stergios Zacharoulis, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No